CLINICAL TRIAL: NCT05398991
Title: A Prospective, Multicenter, Single-arm Trial of Coronary Covered Stents Implantation for the Treatment of Coronary Artery Perforation
Brief Title: Coronary Covered Stents Implantation for the Treatment of Coronary Artery Perforation
Acronym: CONVOY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort Rhythm MedTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-MC-001
Record Dates: First submitted 2022-05-20; First posted 2022-06-01 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Perforation
Keywords: Coronary Artery Perforation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Subjects in experimental group will be implanted with the Coronary Covered Stents System manufactured by Shanghai MicroPort Medical (Group) Co., Ltd.
  Interventions: Device: the Coronary Covered Stents System manufactured by Shanghai MicroPort Medical (Group) Co., Ltd.

INTERVENTIONS:
Device: the Coronary Covered Stents System manufactured by Shanghai MicroPort Medical (Group) Co., Ltd. — the Coronary Covered Stents System contains a covered stent and a delivery system

SUMMARY:
A clinical trial of Coronary Covered Stents System for the treatment of coronary artery perforation.

DETAILED DESCRIPTION:
This is a pre-market clinical investigation aiming to evaluate the safety and effectiveness of Coronary Covered Stents System for the treatment of coronary artery perforation.

ELIGIBILITY:
General Inclusion Criteria

1. Subjects aged ≥ 18 years.
2. Subjects with perforated coronary or aortic-coronary bypass graft vessels.
3. Subjects who are able to understand the purpose of the trial, participate voluntarily or by proxy and indicate by signing the informed consent form that they recognize the risks and benefits described in the informed consent document and are willing to undergo clinical follow-up.

Angiography Inclusion Criteria

1. The lesion is a perforated coronary artery or aortic coronary bypass graft vessel of Ellis type I, type II or type III.
2. Reference vessel diameter from 2.5 mm to 4.0 mm.
3. According to the judgment of the investigator, the perforations require covered stent coverage and for which the covered stent can be delivered.
4. Up to one perforated lesion will be treated and up to one covered stent expected to be implanted.

General Exclusion Criteria

1. Subjects who are unable to receive anticoagulation or antiplatelet therapy.
2. Subjects who are unable to tolerate 6 months of DAPT treatment.
3. Subjects who are allergic to aspirin, heparin, contrast agents, cobalt-based alloys (including metallic elements such as cobalt, chromium, nickel, and tungsten), or polytetrafluoroethylene.
4. According to the judgment of the investigator, subjects who are poorly compliant and unable to complete the study as required; or subjects who are otherwise deemed unsuitable for the enrollment.
5. Primary or secondary cryptogenic coronary perforation or bleeding.
6. Patients who are expected to require treatment with an adjunctive device such as IABP/ECMO.

Angiographic Exclusion Criteria

1. anatomical structures proximal to the target lesion or within the lesion (e.g., severe tortuosity, etc.) that would obstruct delivery of the coronary covered stent.
2. implantation of the covered stent may result in occlusion of a significant coronary branch relevant to the treatment.
3. left or right coronary opening area or coronary sinus entrapment.
4. balloon dilation can not relieve bleeding symptoms
5. Subjects who need to implant two or more covered stents
6. primary or secondary unexplained coronary perforation, or ≥ 2 perforation sites.
7. Other conditions that are not suitable for covered stents treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Procedural Success | During hospitalization (up to 7 days after procedure)
  Successful implantation of a coronary covered stent and sealing of the perforation with ≤30% diameter stenosis(visual inspection) and TIMI III with no blood spillage requiring urgent surgical intervention.

SECONDARY OUTCOMES:
Sealing Success | Index procedure
  No residual blood spillage requiring urgent surgical intervention after successful release of the stent delivery system
Clinical Success | During hospitalization (up to 7 days after procedure)
  on the basis of procedure success with no device-related composite endpoint events during hospitalization (up to 7 days after procedure)
Mortality | 1 month, 6 months, and 1 year postoperatively
  Mortality (Cardiac, cardiovascular, non-cardiovascular)
Myocardial Infarction | 1 month, 6 months, and 1 year postoperatively
  As per Myocardial Infarction (Fourth Universal Definition of Myocardial Infarction) types 1, 2 and 3 MI: have the clinical evidence of acute myocardial ischaemia and with detection of a rise and/or fall of cTn values with at least one value above the 99th percentile URL and at least one of the following:
  * Symptoms of myocardial ischaemia;
  * New ischaemic ECG changes;
  * Development of pathological Q waves;
  * Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality in a pattern consistent with an ischaemic aetiology;
  * Identification of a coronary thrombus by angiography or autopsy (not for types 2 or 3 MIs).
  types 4 and 5 MI: Coronary procedure-related MI ≤ 48 hours after the index procedure is arbitrarily defined by an elevation of cTn values > 5 times for type 4a MI and > 10 times for type 5 MI of the 99th percentile URL in patients with normal baseline values.
Target Lesion Revascularization | 1 month, 6 months, and 1 year postoperatively
  Target Lesion Revascularization (ischemia-driven, non ischemia-driven)
Target Vessel Revascularization | 1 month, 6 months, and 1 year postoperatively
  Target Vessel Revascularization (ischemia-driven, non ischemia-driven)
Rate of emergency surgery or additional pericardial tamponade/puncture postoperatively | 1 month, 6 months, and 1 year postoperatively
  the rate of events caused an emergency surgery, additional pericardial tamponade or puncture postoperatively
Stent thrombosis rate | 1 month, 6 months, and 1 year postoperatively
  s (by Academic Research Consortium [ARC] definitions)
AEs and SAEs | 1 month, 6 months, and 1 year postoperatively
  Adverse Events and Severe Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Qian Tong, M.D., Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No